CLINICAL TRIAL: NCT03918837
Title: Effects of rTMS Over Right COF Blood Perfusion in OCD Patients: an ASL Double Blinded Study
Brief Title: Neurostimulation and OCD, a MRI Study
Acronym: ASLTOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Center Guillaume Régnier (Other)
Collaborators: Fondation de l'Avenir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: RC19_01DD_ASLTOC; 2019-A00165-52 (Other: ANSM)
Record Dates: First submitted 2019-04-11; First posted 2019-04-18 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: Arterial Spin Labeling; Obsessive Compulsive Disorder; Magnetic Resonance Imaging; Repetitive Transcranial Magnetic Stimulation; Double blinded; Sham
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: The investigators will randomize participants between two parallel groups using a randomization list. One group will undergo active rTMS while the second one will undergo sham rTMS. The second group will have the possibility of performing an active rTMS treatment at the end of each patient's participation. All subjects will undergo a MRI with anatomical and ASL sequences one week before treatment and four weeks after treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The masking model will use the same rTMS coil as the active group, bit with a 180° rotation, making the magnetic field face the opposite direction, and thus not being able to produce Neuromodulation on the patient. The stimulation intensity will be decreased at 30% of the motor threshold, to keep the characteristic sound of active rTMS. The patient will not know their group; neither will the investigator nor the rater. Only the rTMS performing technician will know the randomization group to be able to choose the right setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham rTMS (Sham Comparator): The investigators will perform sham rTMS at 30% of the Motor Threshold, with a 1Hz frequency and 1200 pulses during one session. The target will be the right Orbito Frontal Cortex, localized using Neuronavigation. Sessions will last fifteen minutes; subjects will perform two sessions a day during five days. The coil will have a 180° rotation compared to the active coil position, thus making the magnetic field ineffective on the patient's cortex.
  Participants will undergo a MRI with anatomical and ASL sequences one week before and four weeks after treatment.
  All participants of this group will have the opportunity to undergo an active rTMS treatment right after the end of each one's participation in the study.
  Interventions: Other: Sham rTMS
- Active rTMS (Active Comparator): The investigators will perform active rTMS at 120% of the Motor Threshold, with a 1Hz frequency and 1200 pulses during one session. The target will be the right Orbito Frontal Cortex, localized using Neuronavigation. Sessions will last fifteen minutes; subjects will perform two sessions a day during five days.
  Participants will undergo a MRI with anatomical and ASL sequences one week before and four weeks after treatment
  Interventions: Other: Active rTMS

INTERVENTIONS:
Other: Sham rTMS — Participants will undergo sham rTMS for five days with two daily fifteen minutes rTMS sessions.
  Arms: Sham rTMS
Other: Active rTMS — Participants will undergo active rTMS for five days with two daily fifteen minutes rTMS sessions.
  Arms: Active rTMS

SUMMARY:
This study will focus on the use of repetitive Transcranial Magnetic Stimulation (rTMS) as a treatment of Obsessive Compulsive Disorder (OCD), which is a common illness that impairs quality of life and that can be hard to treat.

To precisely analyze the effects of rTMS on OCD, the investigators are going to plan a study comparing cerebral blood flow before and after rTMS treatment. The measuring will occur on the Orbito Frontal Cortex (OFC), whose role in OCD has already been shown by our team (Nauczyciel et al, 2014 in Translational Psychiatry), using Magnetic Resonance Imaging in Arterial Spin Labeling, an MRI method allowing to measure arteriola blood flow.

Our primary outcome is to show a significate difference between cerebral blood flow in OCD between one group of participants treated by rTMS and another one treated by placebo. The study will be double blinded with a placebo rTMS machine, monocentric and prospective, with participants suffering from OCD randomized between two groups.

DETAILED DESCRIPTION:
Obsessive Compulsive Disorders (OCD) are a frequent and debilitating disease. Impact on daily life is usually important, with a high rate of mood and anxious comorbidities, such as Major Depressive Disorder occurring in half of these participants. The effects can be dramatic, leading to higher suicide rate in this population.

Guidelines for OCD treatment in France recommend the use of Serotonin Specific Recapture Inhibitors (SSRI) and Cognitive Behavioral Therapy (CBT), if possible simultaneously. However, those treatments are responsible for adverse effects for the first and not easily accessible for the second. Consequently, a non-negligible number of participants still suffers from symptoms of OCD with a non-optimal treatment.

Repetitive Transcranial Magnetic Stimulation (rTMS), a noninvasive neurostimulation method, has shown its usefulness in the treatment of mental illnesses. It has been authorized by the Food and Drugs Administration in the United States for the treatment of OCD. It represents an alternative method for helping those participants, but pattern of modifications over OCD pathophysiology has still to be unraveled.

In order to precisely analyze the effects of Low Frequency rTMS (LF rTMS) on OCD, the investigators designed a monocentric, prospective, double blind study comparing cerebral blood flow (CBF) before and after a rTMS treatment. Measurements will be performed on the Orbito Frontal Cortex (OFC), whose role in OCD has already been shown by our team (Nauczyciel et al, 2014 in Translational Psychiatry), using Magnetic Resonance Imaging (MRI) in Arterial Spin Labeling (ASL).

Inclusion criteria will be OCD diagnosis, age between 18 and 65, and the lack of counter indication to MRI and rTMS. Participants will firstly undergo MRI before treatment, along with a psychometric assessment. Participants will then receive a one-week rTMS treatment, with two sessions of fifteen minutes per day. Second MRI and evaluation will be performed 4 weeks after the end of the treatment.

Psychometric assessment will consist of MINI, YBOCS, CGI, MADRS, HAMA, and GAF, administered before and four weeks after treatment. The psychiatrist giving the assessment will be blind to the randomization of the patient, so will be the radiologist performing the MRI.

Our primary outcome is to show a significant difference between CBF in OCD in participants treated by rTMS versus participants treated by sham rTMS. A decrease of the CBF in the OFC is expected, in regards to the inhibitor effects of LF rTMS. This result will allow us to follow objectively the neurobiological effects of rTMS, developing the ability to plan more efficiently rTMS treatment for participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants over 18 to 65
* Score at YBOCS over 15
* Diagnosis of Obsessive Compulsive Disorder acknowledged by two psychiatrists using the DSM V criteria
* Patient is able to receive and understand information about the trial, and agrees to participate in the trial
* Indication of treatment by rTMS

Exclusion Criteria:

Related to MRI and / or rTMS:

* Cardiac Stimulator or Implantable Automatic Defibrillator
* Neurosurgical Clips
* Cochlear Implant
* Intra ocular or cranial metallic foreign body
* Endoprosthesis lasting from less than four weeks
* Ostheosynthesis material lasting from less than six weeks
* Claustrophobia

Other criteria:

* Pregnancy or breast feeding
* Unstable hemodynamics, acute respiratory failure, need for constant surveillance not possible during the MRI, precarious general condition
* Patient over legal protection, care without consent
* Active psychiatric pathology other than anxious or mood disorder
* Active severe somatic disease
* History of seizures or other neurologic pathologies (Parkinson's Disease, CVA, Alzheimer's Disease, Multiple Sclerosis, Lewy Body Dementia...)
* Patient without social security

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow of the Orbito-Frontal Cortex from Arterial Spin Labeling Data | one measure four weeks after end of treatment
  Comparison between the sham rTMS group and the active rTMS group will be analyzed from the ASL data about cerebral blood flow in the Orbito-Frontal Cortex. We expect to find a significant difference between the two groups four weeks after the treatment on the mean of cerebral blood flow, as raw data will be converted into numerical data for analysis.

SECONDARY OUTCOMES:
Score at Yale-Brown Obsessive Compulsive Scale (YBOCS) | one measure before treatment, one four weeks after end of treatment
  YBOCS is a scale used to make an accurate and objective measure of the intensity of OCD symptoms for a patient at a precise time, ranging from 0 to 40 (maximum severity), analyzes will be based on each group's mean score.
Score at Montgomery and Asberg Depression Rating Scale (MADRS) | one measure before treatment, one four weeks after end of treatment
  MADRS is a clinical scale used to measure the severity of depressive symptoms for a patient, ranging from 0 to 60 (maximum severity), analyzes will be based on each group's mean score.
Score at General Assessment Functioning Scale (GAF) | one measure before treatment, one four weeks after end of treatment
  GAF is a scale representing the functional abilities of a patient in his daily life and the way his illness potentially impairs his normal social, personal and professional quality of life, ranging from 0 to 100 (representing a normal fully functioning life), analyzes will be based on each group's mean score.
Score at Hamilton Anxiety Rating Scale (HAMA) | one measure before treatment, one four weeks after end of treatment
  HAMA is a scale used to measure the intensity of anxious symptoms of a patient at a given time, ranging from 0 to 60 (maximum severity), analyzes will be based on each group's mean score.
Blindness Evaluation | measure will occur four weeks after the treatment, at the same assessment than clinical outcomes
  Participants will pass an evaluation of their perception of the sham devices, which will allow us to analyze the masking strategy the investigators use considering this double blind study. A five propositions assessment will be used, ranging from 1 to 5 (1 representing the patient's certainty of being in the active treatment group and 5 representing the patient's certainty of being in the sham treatment group). Analyses will be carried using Bang's Blinding Index (Bang et al, Assessment of blinding in clinical trials. Control Clin Trials. 2004).
Intra Group CBF Comparison | one measure before treatment, one four weeks after end of treatment
  We will be using the ASL data to compare the evolution of cerebral blood flow in the Orbito-Frontal Cortex within each patient's brain.
Score at Clinical Global Impression scale (CGI) | one measure before treatment, one four weeks after end of treatment
  CGI is a scale used to give a clinical impression of a patient from the physician's observation, being able to evaluate if the patient's condition has worsened or improved between two evaluations, scores ranging from 0 to 7 (maximum severity or important degradation of the patient's condition), analyzes will be based on each group's mean score.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DRAPIER, MD PHD, Principal Investigator — Centre Hospitalier Guillaume Régnier
Locations (1):
- Centre Hospitalier Guillaume Régnier, Rennes, ille et vilaine, France

IPD SHARING:
Plan to Share IPD: Yes
Data about study protocol and clinical information will be available on request from other researchers. MRI raw data will not be shared but processed data is planned to be available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available from the moment a scientific publication is accepted to 5 years later.
Access Criteria: Access to data will be granted for researchers aiming to perform another analysis or to review the topic, or to perform a meta-analysis.

REFERENCES:
- [Background] Anticevic A, Hu S, Zhang S, Savic A, Billingslea E, Wasylink S, Repovs G, Cole MW, Bednarski S, Krystal JH, Bloch MH, Li CS, Pittenger C. Global resting-state functional magnetic resonance imaging analysis identifies frontal cortex, striatal, and cerebellar dysconnectivity in obsessive-compulsive disorder. Biol Psychiatry. 2014 Apr 15;75(8):595-605. doi: 10.1016/j.biopsych.2013.10.021. Epub 2013 Nov 4. PMID 24314349
- [Background] van der Straten AL, Denys D, van Wingen GA. Impact of treatment on resting cerebral blood flow and metabolism in obsessive compulsive disorder: a meta-analysis. Sci Rep. 2017 Dec 12;7(1):17464. doi: 10.1038/s41598-017-17593-7. PMID 29234089
- [Background] Le Jeune F, Verin M, N'Diaye K, Drapier D, Leray E, Du Montcel ST, Baup N, Pelissolo A, Polosan M, Mallet L, Yelnik J, Devaux B, Fontaine D, Chereau I, Bourguignon A, Peron J, Sauleau P, Raoul S, Garin E, Krebs MO, Jaafari N, Millet B; French Stimulation dans le trouble obsessionnel compulsif (STOC) study group. Decrease of prefrontal metabolism after subthalamic stimulation in obsessive-compulsive disorder: a positron emission tomography study. Biol Psychiatry. 2010 Dec 1;68(11):1016-22. doi: 10.1016/j.biopsych.2010.06.033. Epub 2010 Oct 16. PMID 20951978
- [Background] Nauczyciel C, Le Jeune F, Naudet F, Douabin S, Esquevin A, Verin M, Dondaine T, Robert G, Drapier D, Millet B. Repetitive transcranial magnetic stimulation over the orbitofrontal cortex for obsessive-compulsive disorder: a double-blind, crossover study. Transl Psychiatry. 2014 Sep 9;4(9):e436. doi: 10.1038/tp.2014.62. PMID 25203167
- [Background] Ruffini C, Locatelli M, Lucca A, Benedetti F, Insacco C, Smeraldi E. Augmentation effect of repetitive transcranial magnetic stimulation over the orbitofrontal cortex in drug-resistant obsessive-compulsive disorder patients: a controlled investigation. Prim Care Companion J Clin Psychiatry. 2009;11(5):226-30. doi: 10.4088/PCC.08m00663. PMID 19956460